CLINICAL TRIAL: NCT05037617
Title: The REDUCED-I Pilot Trial: REDucing the Utilization of CEsarean Sections With Induction
Acronym: (REDUCED-I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Stephen Wood, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB21-0614
Record Dates: First submitted 2021-08-19; First posted 2021-09-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Induced; Birth
Keywords: Obstetric Labor Complications; Cesarean section; Induced labour; oxytocin
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Dilatation; Oxytocin

STUDY DESIGN:
Intervention Model Description: Once a patient is found to be >=6 cm dilation, the patient will received a blinded vial of oxytocin or saline, which will be numbered according to the random allocation sequence created by the study statistician.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once a patient is found to be ≥6 cm dilation, the study medication will be initiated. Pharmacy will make up identical vials of oxytocin or saline, which will be numbered according to the random allocation sequence created by the study statistician. Nurses will use the blinded vials for ongoing infusion. Patients and caregivers will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention site (Foothills Medical Centre): Continuation of Oxytocin (Experimental): Participants in this arm will receive a blinded vial of oxytocin once a patient is found to be >= 6 cm dilated.
  Interventions: Drug: Continuation or discontinuation of oxytocin during the active first stage of labor (≥6 cm dilation).
- Intervention site (Foothills Medical Centre): Discontinuation of oxytocin (Placebo Comparator): Participants in this arm will receive a blinded vial of saline solution once a patient is found to be >= 6 cm dilated.
  Interventions: Drug: Continuation or discontinuation of oxytocin during the active first stage of labor (≥6 cm dilation).

INTERVENTIONS:
Drug: Continuation or discontinuation of oxytocin during the active first stage of labor (≥6 cm dilation). — At the intervention site (Foothills Medical Centre), for participants who consent to being part of the trial, once a patient is found to be >= 6 cm dilation, the study medication will be initiated. Pharmacy will make up identical vials of oxytocin or saline, which will be numbered according to the random allocation sequence created by the study statistician.
  The intervention will be continued until delivery unless contractions decrease to less than 2 in 10 minutes or if no further cervical dilation is noted 4 hours after discontinuation.
  Other Names: oxytocin

SUMMARY:
This pilot project is a randomized controlled trial where induced patients receive an intervention of oxytocin discontinuation once in the active stage of labor (≥6 cm dilation). The intent is to reduce uterine hyperstimulation and fetal distress, therefore, lowering cesarean sections (CS) in first time mothers at term (≥ 37 weeks), with a cephalic presenting singleton fetus, without increasing maternal or neonatal morbidity. If REDUCE-I pilot trial suggests a safe reduction in CS rates and patient satisfaction, application for a multi-centre randomized controlled trial would follow.

DETAILED DESCRIPTION:
This pilot project is a randomized controlled trial of a proposed intervention to modify management of labor inductions once in the active first stage of labor. The intervention will take place at Foothills Medical Centre (FMC). Randomization will be computer generated, participants will be stratified by need for cervical ripening and randomization will be blocked. Participants will be primiparous women 18 years old or older, at term (≥ 37 weeks) with a cephalic presenting singelton fetus undergoing induction of labor with oxytocin. Once patients are in the active first stage of labor, study medication will be initiated (identical vials of oxytocin or saline prepared by the Alberta Health Services Research Pharmacy). Treatment period will continue until delivery. If the frequency of contractions are reduced to less than 2 in 10 minutes or there has been no change in dilation for 4 hours, then oxytocin can be restarted.

Royal Alexandra Hospital in Edmonton will be used as a contemporaneous non-intervention control site.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women undergoing induction of labor with oxytocin.
* Primiparous
* 18 years old or older
* at term (≥37 weeks)
* cephalic presenting
* singleton fetus

Exclusion Criteria:

* Multiple pregnancies
* known fetal congenital or chromosomal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Rate of Cesarean section in labor | At Delivery
  Rate of Cesarean section in labor
Occurrence of Uterine Hyperstimulation | During labour, after >=6 cm dilation
  Occurrence of >5 contractions in 10 minutes
Proportion of screened subjects who agree to enroll in the trial | During screening of potential participants
  Proportion of screened subjects who agree to enroll in the trial

SECONDARY OUTCOMES:
Rate of perinatal death | At delivery
  Rate of perinatal death
Rate of neonatal asphyxia | At delivery
  Neonatal asphyxia is defined as intrapartum stillbirth or neonatal death from asphyxia (Perinatal Society of Australia and New Zealand coding) or Neonatal Intensive Care Unit admission and at least two of: a. Apgar score of ≤5 at 10 minutes; b. Mechanical ventilation or chest compressions for resuscitation within 10 minutes; c. Cord pH < 7.00 (venous or arterial), or arterial base excess ≥ 12 at birth. Rate of neonatal asphyxia for deliveries involving primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of moderate or severe asphyxia (Sarnat) or meets criteria for therapeutic cooling | At delivery
  Rate of moderate or severe asphyxia (Sarnat) or meets criteria for therapeutic cooling
Rate of neonatal sepsis or suspected sepsis | At delivery
  Rate of neonatal sepsis or suspected sepsis
Rate of postpartum hemorrhage | At delivery
  Rate of postpartum hemorrhage
Rate of blood transfusion | At delivery
  Rate of blood transfusion
Rate of postpartum uterine artery/pelvic artery embolization | Within 28 days of delivery
  Rate of postpartum uterine artery/pelvic artery embolization
Rate of postpartum hysterectomy | Within 28 days of delivery
  Rate of postpartum hysterectomy
Rate of postpartum maternal intensive care unit (ICU) admission | At delivery
  Rate of postpartum maternal intensive care unit (ICU) admission

OTHER OUTCOMES:
Duration of oxytocin discontinuation | During labour, after >=6 cm dilation
  Duration of oxytocin discontinuation
Rate of reintroduction of oxytocin infusion | During labour, after >=6 cm dilation
  Rate of reintroduction of oxytocin infusion

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Wood, MD, FRCSC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT05037617/Prot_SAP_003.pdf